CLINICAL TRIAL: NCT07165574
Title: Prevalence of Anticholinergics in Geriatric Patients With Acute Functional Deterioration
Status: Not yet recruiting | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Riis, MD, Aalborg University Hospital
Other Study IDs: 1-45-72-442-25
Record Dates: First submitted 2025-08-28; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Frailty in Older Adults; Functional Decline; Anticholinergic Syndrome
MeSH Terms: conditions — Anticholinergic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention as the study is observational — As this is an observation study, participants are not assigned an intervention as part of the study

SUMMARY:
This study investigates the anticholinergic burden on patients seen in the Subacute mobile outpatient geriatric clinic in Aalborg, Denmark, between the years of 2024 and 2025.

The age demographic in Denmark and multiple other countries is changing rapidly, with more old and very old individuals as a result. As humans become older, they tend to accumulate more illnesses, and the risk of polypharmacy increases. There is a wide selection of medicine that affect the binding of acetylcholine to the muscarinic receptors, which is either the intended function of the pharmacological product or a side effect.

Since there is no built-in feature in computer systems used by doctors to calculate the cumulative anticholinergic burden, it is often not recognized, thus not reflected upon.

This raises concerns about potential central and peripheral side effects, such as altered mental status, visual disturbances, tachycardia, urinary and fecal retention, dry skin etc.

The study aims to determine the prevalence of anticholinergics in the last 100 patients seen by the Subacute mobile outpatient geriatric clinic in Aalborg University Hospital. The patients are placed in municipal extended-care facilities. Furthermore, the study will investigate the prevalence of anticholinergic side effects concerning the burden on this population.

The study is a retrospective chart review of patient charts from the years of 2024 and 2025, analyzing patient characteristics, comorbidities, medication lists, and calculating the anticholinergic burden through the ACB calculator.

ELIGIBILITY:
Inclusion Criteria:

* patients seen by the Subacute outpatient geriatric clinic at Aalborg University hospital, Denmark, between 2024 and 2025.
* Consecutive sampling starting with the most recent patient chart and going backwards.
* Inclusion is based on chart review and all patients are therefore included consecutively.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient seen by the subactue outpatient geratric clinic at Aalborg University Hospital are older adults who have experienced an acute deterioration of daily function, usually due to acute illness and are admittet to municipality reablement services with the goal of postacute rehabilitation to previous funciton and avoiding nursing home admission. Patients may have been recently discharged from hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anticholinergics | Day 1. That is on the day of patients first contact with the subacute outpatient geratric function at Aalborg Unviversity Hospital
  Number of patients taking anticholinercis (yes/no) defined by the Anticholingeric Cognitive Burden scale (any score above 0)

SECONDARY OUTCOMES:
Prevalence of central side effects | On the day of patients first contact with the subacute outpatient geratric function at Aalborg Unviversity Hospital
  Prevalence of any of the following conditions as described in patient charts: Delirium, other confusion, restlessness, hallucinations, Amnesia, dysarthria, ataxia, stupor, coma.
Prevalence of peripheral anticholinergic side effects | On the day of patients first contact with the subacute outpatient geratric function at Aalborg Unviversity Hospital
  Prevalence of any of the following conditions as described in patient charts: Urinary retention, constipation, tachycardia, visual disturbances, dry skin, dry mouth.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatric Medicine, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided